CLINICAL TRIAL: NCT05212818
Title: A Phase 2, Multicenter, Randomized, Double-blind (Within Dose), Placebo-controlled, Parallel-group, and Dose-range-finding to Evaluate the Efficacy and Safety in Treatments for COVID-19 in Hospitalized Adults
Brief Title: Evaluate the Efficacy and Safety of TF0023 in Treatments for COVID-19 in Hospitalized Adults
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low patient accrual.
Sponsor: Techfields Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TF-TF0023-201
Record Dates: First submitted 2022-01-20; First posted 2022-01-28 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: COVID-19 Pneumonia
Keywords: Pneumonia; COVID-19
MeSH Terms: conditions — Pneumonia; COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Low Dose of Active Drug (Experimental): 80 patients will be randomly assigned to low dose, take active drug BID.
  Interventions: Drug: TF0023
- Low Dose Placebo Control (Experimental): 80 patients will be randomly assigned to Low dose placebo, take the placebo BID.
  Interventions: Drug: TF0023
- High Dose of Active Drug (Experimental): 160 patients will be randomly assigned to high dose, take the active drug BID.
  Interventions: Drug: TF0023
- High Dose Placebo Control (Experimental): 80 will be randomly assigned to high dose placebo, take the placebo BID.
  Interventions: Drug: TF0023

INTERVENTIONS:
Drug: TF0023 — Techfields Inc. is developing TF0023, a new investigational prodrug, indicated for relief of the signs and symptoms of ARDS and pneumonia caused by COVID-19 and other viruses.
  Other Names: IP, Active drug

SUMMARY:
Techfields Inc. is developing a new investigational prodrug as a topical spray, indicated for relief of the signs and symptoms of ARDS and pneumonia caused by COVID-19. This is a Phase 2, Multicenter, Randomized, Double-blind (Within Dose), Placebo-controlled, Parallel-group, and Dose-range-finding Study to Evaluate the Efficacy and Safety of Active drug Versus Placebo in Treatments for COVID-19 in Hospitalized Adults, relieving of the signs and symptoms of acute respiratory distress syndrome (ARDS) and pneumonia caused by coronavirus disease 2019 (COVID-19).

DETAILED DESCRIPTION:
A total of approximately 400 eligible patients will be randomly assigned to receive Active Drug low dose (n=80), placebo low dose (n=80), Active Drug high dose (n=160), or placebo high dose (n=80) according to a 1:1:2:1 ratio. The study will be stopped when the last patient completes the double-blind treatment period (end of treatment [EOT]/early termination visit [ETV] on Day 29 + 3 days) and follow-up period. Screening will start when the patient is hospitalized. Each patient enrolled will receive an investigational product (IP; Active Drug or placebo) in a double-blind manner for 28 days (during the double-blind treatment period), starting immediately after all eligibility criteria (including test results) are confirmed. All patients will receive institutional standard of care (SOC) concurrently with their assigned IP. There will be a follow-up visit on Day 36+3 days.

ELIGIBILITY:
Inclusion Criteria:

1. Admitted to a hospital with pulmonary symptoms of active COVID-19.
2. Patient (or legally authorized representative) provides informed consent prior to initiation of any study procedures.
3. Patient (or legally authorized representative) understands and agrees to comply with planned study procedures.
4. Male or nonpregnant female adult ≥18 years of age at time of enrollment.
5. Has laboratory confirmed severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection as determined by polymerase chain reaction (PCR) or other commercial or public health assay (serology is not acceptable) in any specimen, as documented by either of the following:

   1. Laboratory confirmed SARS-CoV-2 infection by method as defined above, in sample collected <72 hours prior to randomization; OR
   2. Laboratory confirmed SARS-CoV-2 infection by method as defined above, in sample collected ≥72 hours prior to randomization, documented inability to obtain a repeat sample (e.g., due to lack of testing supplies, limited testing capacity, results taking >24 hours, etc.) AND progressive disease suggestive of ongoing SARS-CoV-2 infection.
6. Has a score of 4 (hospitalized, oxygen by mask or nasal prongs), 5 (hospitalized, noninvasive ventilation or high-flow oxygen), or 6 (hospitalized, intubation and mechanical ventilation) in the ordinal scale.
7. Women of childbearing potential must agree to either abstinence or use at least 1 primary form of contraception not including hormonal contraception from the time of screening through Day 29. (Double-barrier method [condoms, sponge, diaphragm, with spermicidal jellies, or cream] is acceptable).
8. Agrees to not participate in another clinical study for the treatment of COVID-19 or SARS-CoV-2 through Day 29. However, Food and Drug Administration (FDA)-approved or under an emergency use authorization antivirus or other drugs may be allowed, and that should be judged by the patient's physician.

Exclusion Criteria:

1. Any condition, including any significant medical or neuropsychiatric condition, including the presence of laboratory abnormalities, which in the judgment of the investigator places the patient at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study including, but not limited to:

   1. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >3 × the upper limit of normal (ULN) at screening.
   2. Total bilirubin or alkaline phosphatase level >3.0 × the ULN at screening.
   3. Platelet count <100 × 109/L.
2. Extracorporeal membrane oxygenation required at baseline.
3. Stage 3 or end stage renal disease (ESRD) patients with acute renal insufficiency may be considered only after discussion with medical monitor.
4. Is at increased risk for bleeding events (e.g., had recent cerebral hemorrhage, gastrointestinal bleeding, serious trauma, recent surgery, or organ biopsy).
5. Pregnant (patient has a positive pregnancy test result at screening) or breast-feeding.
6. Anticipated discharge from the hospital or transfer to another hospital which is not a study site.
7. Allergy to any study medication or known allergy to nonsteroidal anti-inflammatory drugs, including aspirin.
8. Patient must agree to refrain from taking oral aspirin or any orally administered acetylsalicylic acid medications until PK sampling is completed to be eligible to participate in the PK sub-study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-03-08 (Actual)

PRIMARY OUTCOMES:
Percentage of patients able to maintain peripheral capillary oxygen saturation (SpO2) of >93% without oxygen support at Day 15. | 15 days
  To evaluate the clinical efficacy of Active drug relative to the control arm in patients hospitalized with respiratory impairment from acute COVID-19 as assessed by the ability to maintain peripheral capillary oxygen saturation (SpO2) of >93% without supplemental oxygen.

SECONDARY OUTCOMES:
Time to not requiring oxygen support. | 28 days
  To evaluate the clinical effect of Active drug as compared to placebo, as assessed by time to not require supplemental oxygen.
Cumulative incidence of SAEs, Grade 3 and 4 clinical and/or laboratory AEs | 28 days
  To evaluate the safety of Active drug compared to placebo.
Changes of clinical status (9-point ordinal scale) | 15 days
  To evaluate the clinical efficacy of Active drug as compared to placebo, as assessed by clinical status (9-point ordinal scale) at Day 15.
Number of supplemental oxygen-free days between Day 1 and Day 29. | 28 days
  To evaluate the clinical effect of Active drug compared to placebo, as assessed by supplemental oxygen requirements, and oxygenation.
Changes of chest x-ray, and computerized tomography (CT) scan | 28 days
  To evaluate the clinical effect of Active drug compared to placebo as assessed by chest x-ray, and computerized tomography (CT) scan.
Changes of clinical status (9-point ordinal scale) | 28 days
  To evaluate the clinical efficacy of Active drug as compared to placebo, as assessed by clinical status (9-point ordinal scale) at Day 15.
Percentage of patients reporting each severity rating on the 9-point ordinal scale | 28 days
  To evaluate the efficacy of Active drug compared to placebo as assessed by percentage of patients reporting each severity rating on the 9-point ordinal scale.
All-cause mortality | 28 days
  To evaluate the efficacy of Active drug compared to placebo on all-cause mortality (ACM).
Pattern score and volumetric score of the radiologic severity index. | 28 days
  To evaluate the efficacy of Active drug compared to placebo as assessed by pattern score and volumetric score of the radiologic severity index.
Duration of hospitalization and duration of Intensive Care Unit (ICU) treatment | 28 days
  To evaluate the efficacy of Active drug compared to placebo for patient clinical status on duration of hospitalization and duration of Intensive Care Unit (ICU) treatment.
Incidence and duration of new mechanical ventilation use and on respiratory failure-free days | 28 days
  To evaluate the efficacy of Active drug compared to placebo for patient clinical status on incidence and duration of new mechanical ventilation use and on respiratory failure-free days.

CONTACTS AND LOCATIONS:
Overall Officials: Chongxi Yu, Ph.D, Study Chair — Techfields Inc
Locations (5):
- United States (3):
  - White Oak Medical Center LLC, Gaithersburg, Maryland
  - Holy Name Medical Center, Teaneck, New Jersey
  - Lincoln Medical Center, The Bronx, New York
- South Africa (2):
  - Worthwhile Clinical Trial, Benoni, Gauteng
  - Dr JM Engelbrecht Trials Site, Somerset West, Western Cape

IPD SHARING:
Plan to Share IPD: No